CLINICAL TRIAL: NCT05357729
Title: Safety and Performance Study of the MultiSense® Ambulatory Telemonitoring System for Non-critical Patient Management
Acronym: TELESENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Collaborators: Rhythm Diagnostic Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-004
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Visceral and Digestive Surgery; Post-surgical Monitoring; Post-surgical Rehabilitation
Keywords: Vital signs; Connected device; real-time monitoring; post-surgery monitoring; cardio-respiratory monitoring; telemonitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MultiSense® remote monitoring (Experimental): The patients included will be equipped with the MultiSense® solution prior to the hospital discharge. The device will be used for 6 days from the date of actual deployment.
  Interventions: Device: MultiSense® remote monitoring

INTERVENTIONS:
Device: MultiSense® remote monitoring — At hospital, the patient will be monitored with conventional monitoring devices as well as the MultiSense® solution (at least one hour with a reference monitor). After hospital discharge, the patients will be remotely monitored by their healthcare professional using the MultiSense® solution.

SUMMARY:
In this clinical investigation, the investigators will assess the safety, performances and clinical added value of the MultiSense® ambulatory telemonitoring solution in real-life situations.

DETAILED DESCRIPTION:
The MultiSense® solution is a medical device for telemonitoring for in and outpatient use.

It includes 5 physiological data sensors and communicates via Bluetooth with a smartphone. The data is centralized in the web and a web application allows healthcare professionals to scrutinize patient's data.

Among its potential benefits, the MultiSense® solution offers continuous, non-invasive and wireless physiological data recording over 5 days whenever patient monitoring is needed. There is a special focus on the post-operative monitoring, especially during the initial convalescence phase outside the hospital. An automatic notification system can be set up by a healthcare professional to notify abnormal data and potential need for phone call and/or physical home intervention.

The aim of this study is to evaluate the safety, the performance and added value of the MultiSense® solution in real-life situations. The study population includes 20 post-surgical patients having a genuine need for post-hospital monitoring and be likely to have variations in physiological variables monitored, without being in a critical condition. The patients included will be equipped with the MultiSense® solution prior to the hospital discharge. The device will be used for 6 days from the date of actual deployment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (male or female over 18 years) in non-critical care settings
2. Patient programmed for an elective surgery
3. Need to monitor at home at least one physiological parameter: heart rate, respiratory rate, SpO2, temperature, physical activity
4. Patient able to use a smartphone
5. Patient with Wi-Fi and/or Cellular connectivity at home
6. Patient with a personal phone which allows to receive text messages
7. Patient able to receive and understand information related to the study and give written informed consent
8. Patient affiliated to the French social security system

Exclusion Criteria:

1. Patient with known skin allergy (adhesive or silicon) or skin disease that would not allow the use of an adhesive
2. Patient with an active implantable device (such as a pacemaker or automatic defibrillator)
3. Patient with an elective imagery planned during the use of MultiSense
4. Pregnant or lactating patient
5. Patient in exclusion period (determined by a previous or a current study)
6. Patient under guardianship or trusteeship
7. Patient under the protection of justice or deprived of liberty
8. Patient in situation of emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Determination of the safety and performance of the MultiSense® solution in patient monitoring, in terms of heart rate accuracy by comparison with a reference monitor. | From patch placement to hospital discharge, assessed up to 3 hours
  Accuracy is defined as an average measurement variation less than 5 bpm of the mean value, with respect to the reference standard
Determination of the safety and performance of the MultiSense® solution in patient monitoring, in terms of data availability. | From patch placement to removal, assessed up to 7 days
  Percentage of missing data due to technical issues (non-behavioral events) over the monitoring period below 15%.
Determination of the safety and performance of the MultiSense® solution in patient monitoring, in terms of data artefacts. | From patch placement to removal, assessed up to 7 days
  Percentage of artefacts due to technical issues (non-behavioral events) over the monitoring period below 10% for heart rate, 20% for the respiratory rate or 30% for SpO2.
Determination of the safety and performance of the MultiSense® solution in patient monitoring, in terms of data transmission. | From patch placement to removal, assessed up to 7 days
  Data transmission is defined as more than 90% of data with transmission time from patch to server less than 5 min.

SECONDARY OUTCOMES:
Patient's tolerance to prolonged use of the MultiSense® solution (Safety in use, side effects) | From patch placement to its removal (up to 7 days)
  Accounting and classification of unexpected local and distant event due to the use of the MultiSense® solution (vigilance data) and Patient's questionnaire
Device defects | From patch placement to its removal (up to 7 days)
  Accounting of device deficiencies reported by the investigator, the patient or identified by MultiSense data analysis
Clinical relevance of the notifications provided by MultiSense® solution | From patch placement to its removal (up to 7 days)
  Relevance of the notifications generated by MultiSense® will be judged on the relevance of the notification's functionality by the healthcare professional in real-life situation by the mean of a questionnaire (4-levels Likert scale)
Clinical relevance of the notifications provided by MultiSense® solution | From patch placement to its removal (up to 7 days)
  Relevance of the notifications generated by MultiSense® will be judged on the relevance of the notification's functionality by the healthcare professional in real-life situation by the mean of notification treatment through MultiSense® web application
Remote monitoring facilitation for the healthcare professional through the solution's ease of use and satisfaction gained | From patch placement to its removal (up to 7 days)
  Determination of healthcare professionals' practical interest in the solution and satisfaction of use assessed via a questionnaire (4-levels Likert scale)
Patient's satisfaction and reassurance when monitored by the device | From patch placement to its removal (up to 7 days)
  Determination of patient satisfaction and reassurance by an end-study questionnaire (4-levels Likert scale)
Patch autonomy | From patch placement to its removal (up to 7 days)
  Percentage of patches with an autonomy > 5 days including skin adhesion and battery life (MultiSense® data and patient's questionnaire)
Respiratory rate accuracy in terms of impedance | From patch placement to hospital discharge, assessed up to 3 hours
  Respiratory rate accuracy by comparison of MultiSense® data with the reference monitor in terms of impedance
Respiratory rate accuracy in terms of EtCO2 | From patch placement to hospital discharge, assessed up to 3 hours
  Respiratory rate accuracy by comparison of MultiSense® data with the reference monitor in terms of EtCO2
Estimation of posture and activity level reported by the MultiSense® solution | From patch placement to its removal (up to 7 days)
  Determination of the posture and activity level consistency by accounting the percentage of lying position and low activity at night and the percentage of high activity during day (MultiSense® data)
MultiSense® data quality after moderate level of activity | From patch placement to its removal (up to 7 days)
  Distribution of activity level across monitoring period, number of showers taken over the monitoring period and evolution of the artefact's metric (as defined in the primary endpoint) over time (MultiSense® data)
Correlation between body temperature and skin temperature | From patch placement to hospital discharge, assessed up to 2 days
  Correlation between the body temperature measured with a standard device and the skin temperature measured with the MultiSense® solution
End of study hardware recovery rate | From patch removal to material return, assessed up to 1 month
  Percentage of MultiSense® patch and gateway returned to RDS at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Michel VIX, MD, Principal Investigator — Service de Chirurgie Digestive, NHC, HUS
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No